CLINICAL TRIAL: NCT06069271
Title: The Immediate Effects of a Standardized Kettlebell Swing Protocol on Lumbar Paraspinal Muscle Function
Brief Title: Kettlebell Swings and Paraspinal Muscle Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Responsible Party: Principal Investigator, Randi Richardson, Clinical Assistant Professor, University of Central Florida
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00001277
Record Dates: First submitted 2023-09-25; First posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Exercise Training

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Who Masked: Outcomes Assessor
Masking Description: Assessor was blinded to group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rest (No Intervention): Subjects in the control group were instructed to complete the general warm up followed by a 10-minute rest period.
- Exercise (Experimental): The intervention group completed two-handed Russian KBSs using an interval training protocol outlined by Jay et al.10 involving 30 seconds of work followed by 30 seconds of rest for 10 total intervals. Prior to completing the intervention, participants completed a general warmup consisting of 10 non-weighted squats, 10 non-weighted dead-lifts, and 10 dowel rod shoulder flexion repetitions. Participants were instructed to perform all warm-up activities at an intensity of 70% of maximal effort using a Rate of Perceived Exertion scale(RPE).
  Interventions: Other: Kettlebell swing

INTERVENTIONS:
Other: Kettlebell swing — The intervention group completed two-handed Russian KBSs using an interval training protocol outlined by Jay et al.10 involving 30 seconds of work followed by 30 seconds of rest for 10 total intervals. Prior to completing the intervention, participants completed a general warmup consisting of 10 non-weighted squats, 10 non-weighted dead-lifts, and 10 dowel rod shoulder flexion repetitions. Participants were instructed to perform all warm-up activities at an intensity of 70% of maximal effort using a Rate of Perceived Exertion scale(RPE).
  Arms: Exercise

SUMMARY:
The purpose of this randomized control trial is to determine the extent of muscle fatigue in the lumbar erector spinae musculature secondary to a high-intensity interval kettlebell swing protocol utilizing TMG previously published by Jay et. al in 2011.

DETAILED DESCRIPTION:
Background: Kettlebell swings are commonly utilized to target the lumbar erector spinae and lower body musculature. This exercise exhibits distinct loading properties that requires cyclical contraction of the trunk extensors and posterior chain, potentially explaining its novel influence on muscle contractility. Tensiomyography (TMG) is a reliable, noninvasive, passive technique that may be used to examine muscular fatigue produced by kettlebell swings. Purpose: The purpose of this randomized control trial is to determine the extent of muscle fatigue in the lumbar erector spinae musculature secondary to a high-intensity interval kettlebell swing protocol utilizing TMG previously published by Jay et. al in 2011. Subjects: Forty-one adults between the ages of 18 and 45 were recruited. Inclusion criteria included subjects with no recent history of low back pain and clearance by the physical activity readiness questionnaire. Methods: Participants were randomly allocated to either a kettlebell swing group (KBS; n=21) or a control group (CON; n=20) who only performed the unloaded warm up. Participants were assessed at baseline, post-intervention, and 24-hours post-intervention for bilateral erector spinae fatigue, measured by five TMG parameters (Dm, Tc, Tr, Td, Ts).

ELIGIBILITY:
Inclusion Criteria:

* Ages of 18 and 45 years of age.
* Clear PAR-Q

Exclusion Criteria:

* history of low back pain
* pre-existing injuries
* If "YES" was the response to any of the seven questions in the PAR-Q, the participant was deemed to be unable to exercise safely.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2020-03-04 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Tensiomyography | Baseline, immediate after exercise, 24 hours after exercise
  Research has progressed to support the test-retest and inter-rater reliability using TMG for measurement of muscle contraction. TMG demonstrates good to excellent relative reliability(0.80-0.99) and inter-rater ICC between 0.77-0.97 Across all five TMG parameters.4-7

CONTACTS AND LOCATIONS:
Overall Officials: William J Hanney, PhD, Study Director — University of Central Florida
Locations (1):
- University of Central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hanney WJ, Perez A, Collado G, Palmer AC, Wilson AT, Richardson RM, Kolber MJ. The Immediate Effects of a Standardized Kettlebell Swing Protocol on Lumbar Paraspinal Muscle Function: A Randomized Controlled Trial. J Strength Cond Res. 2024 Nov 1;38(11):1854-1859. doi: 10.1519/JSC.0000000000004892. Epub 2024 Aug 14. PMID 39178062